CLINICAL TRIAL: NCT06847698
Title: Phase 1, Double-Blinded, Placebo-Controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Safety and Pharmacokinetics Trial of AVR-48
Brief Title: Single Ascending Dose and Multiple Ascending Dose Study of AVR-48
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AyuVis Research, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: AVR-48-01-001
Record Dates: First submitted 2024-08-27; First posted 2025-02-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Safety Issues; Tolerability; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Intervention Model Description: Part A: Eight (8) subjects will participate in each of the 3 dose groups. Subjects will be randomized to receive either AVR-48 or placebo by IV (6 active, 2 placebo per group of 8).
  Part B: Eight (8) subjects will participate in each of the 3 dose groups. Subjects will be randomized to receive either AVR-48 or placebo by IV (6 active, 2 placebo per group of 8).
Who Masked: Participant, Investigator
Masking Description: The investigators, study coordinators, study subjects and the Sponsor will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug: AVR-48 (Experimental): AVR-48 is a small molecule with TLR4 modulating activity and macrophage modulator
  Interventions: Drug: AVR-48
- Drug: Placebo (Placebo Comparator): 0.9% saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVR-48 — Investigational drug reconstituted in normal saline will be administered via IV
  Arms: Drug: AVR-48
Drug: Placebo — Normal saline will be administered via IV
  Arms: Drug: Placebo

SUMMARY:
This is a Phase 1 (healthy adult volunteers), 2-part, double-blind, randomized, placebo controlled trial to evaluate the safety and pharmacokinetic (PK) profiles of escalating single doses of AVR-48 versus placebo (SAD) and escalating multiple doses of AVR-48 versus placebo (MAD). SAD will be initiated first and include a sentinel dosing design. MAD will not utilize a sentinel design unless the safety monitoring committee requests the addition of sentinels. The MAD will be initiated once the lowest doses from SAD are deemed safe.

DETAILED DESCRIPTION:
This is a Phase 1, 2-part, double-blinded, placebo-controlled, randomized SAD/MAD study.

The study will include 2 parts:

* Part A: SAD phase
* Part B: MAD phase

Part A - SAD phase Healthy adult subjects will be randomized to receive a single IV dose of either AVR-48 or placebo in each of 3 planned SAD cohorts. Each cohort will consist of 8 subjects in a 3:1 (active:placebo) ratio to have a total of 6 subjects receiving AVR-48 and 2 subjects receiving placebo. Each cohort will be comprised of 50% male and 50% female subjects.

All SAD cohorts will be dosed according to a sentinel dosing design to ensure safety. Initially, 2 subjects will be dosed; 1 subject will be dosed with AVR-48 and 1 subject with placebo. Blood samples for PK and safety clinical laboratory tests will be collected over the following 24 hours. If the site Principal Investigator (PI), in conjunction with the AyuVis sponsored Independent Medical Monitor, determines that acceptable safety is observed in the sentinel administration, the remaining subjects in the cohort will be dosed and identical safety and PK procedures will be performed; 5 subjects will be dosed with AVR-48 and 1 subject with placebo. Sentinel subjects will be dosed at least 48 hours prior to enrolling the remaining subjects of the cohort. All subjects will be followed for 48 hours post-dose.

Blood samples will be collected periodically for PK, cytokine panels, metabolite assessment, and safety labs; urine samples will be collected periodically for metabolite assessment, and routine safety assessments will be completed daily.

Escalation to the next higher dose will only proceed if none of the stopping criteria have been reached and when the safety and tolerability and available plasma PK analysis of the previous dose are acceptable to the site PI, Sponsor, and Safety Monitoring Committee (SMC). A minimum of 3 days will separate each dose escalation.

Part B - MAD phase Healthy adult subjects will be randomized to receive multiple IV doses of either AVR-48 or placebo in each of 3 planned MAD cohorts. Each cohort will consist of 8 subjects in a 3:1 (active: placebo) ratio to have a total of 6 subjects receiving AVR-48 and 2 subjects receiving placebo. A balance of male and female subjects in each cohort will be attempted, but the final ratio of subject sex will be determined by the available subjects who pass screening at the time of enrollment.

For Cohort 1 and Cohort 2, AVR-48 or matching placebo will be administered twice daily, every 12 hours, for a total of 13 doses over 7 days. For Cohort 3, AVR-48 will be administered once daily, for a total of 7 doses over 7 days. Subjects will be monitored for 48 hours after the last dose and will attend a follow-up visit 7 days after dosing completes.

Blood samples will be collected periodically for PK, cytokine panels, metabolite assessment, and safety labs; urine samples will be collected periodically for metabolite assessment, and routine safety assessments will be completed daily.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF).
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Healthy adult male or female, aged 18 to 55, inclusive, at Screening.
4. Continuous non smoker who has not used nicotine containing products (including e- vaping) for at least 3 months prior to the first dosing and throughout the study
5. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening, and a minimum weight of at least 50.0 kg and a maximum weight of 100.0 kg at screening.
6. Medically healthy with no clinically significant abnormalities in medical history, physical and neurologic examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
7. If female of childbearing potential, must be consistently using an effective method of contraception from screening visit until 30 days after the last drug administration.
8. If female and not of childbearing potential, must be either surgically sterile or post menopausal (i.e., more than 1 year since last menstrual period).
9. A non-vasectomized, male subject must agree to use an effective method of birth control with female partners of childbearing potential during the study and to refrain from donating sperm for 90 days following dosing.
10. No restrictions are required for a vasectomized male subject provided his vasectomy has been performed 4 months or more (and have official documentation) prior to Study Day 1. A subject who has been vasectomized less than 4 months prior to Study Day 1 or does not have official documentation of his vasectomy must follow the same restrictions as a non-vasectomized subject.

Exclusion Criteria:

1. Are mentally or legally incapacitated or have significant emotional problems at the time of the screening visit or expected during the conduct of the study in the opinion of the PI or designee.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
5. Has had surgery or any medical condition within 6 months prior to first dosing which may affect the distribution, metabolism, or elimination of the study drug, in the opinion of the PI or designee.
6. Female subjects with a positive pregnancy test or who are lactating.
7. Positive urine drug or alcohol results at screening or first check-in.
8. Positive cotinine results at screening.
9. Positive result at screening for tuberculosis (i.e., positive result for QuantiFERON TB-Gold).
10. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
11. Unable to refrain from or anticipates the use of:

    • Any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing and throughout the study. After first dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee. Hormone replacement therapy will be allowed.
12. Donation or loss of 50 to 499 mL whole blood within 30 days or more than 499 mL whole blood within 56 days prior to the first dosing.
13. Plasma donation within 14 days prior to the first dosing.
14. Participation in another clinical study within 30 days prior to the first dosing. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.
15. Had a treatment with other investigational drug within 5 times the terminal elimination half-life (t1/2), if known (e.g., a marketed product) or within 30 days (if the t1/2 is unknown), whichever is longer, prior to Study Day 1 dosing.
16. Evidence of Coronavirus Disease 2019 (COVID-19) infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience Adverse Events (AEs), Serious Adverse Events | Up to 16 days
  Number of AEs, SAEs, and discontinuation due to AEs
Number of participants who experience ECG abnormalities | Up to 16 days
  Number of participants with potentially clinically significant ECG readings
Number of participants who experience vital sign abnormalities | Up to 16 days
  Number of participants with potentially clinically significant vital sign values
Number of participants who experience laboratory test abnormalities | Up to 16 days
  Number of participants with potentially clinically significant laboratory test results
Number of participants who experience physical examination abnormalities | Up to 16 days
  Number of participants with potentially significant physical examination findings

SECONDARY OUTCOMES:
PK of AVR-48 in plasma: Area under the plasma-concentration time curve (AUC) | Up to 8 days
  Blood Samples will be collected for plasma analysis
Title: PK of AVR-48 in plasma: Area under the concentration time curve, from time 0 to the last observed non-zero concentration (AUC0-tlast) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Maximum observed concentration (Cmax) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Trough or minimum concentration (Ctrough) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Concentration at the end of the dosing interval (Ct) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Time to maximal observed concentration (tmax) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Accumulation ratio (comparing Day 5 Cmax to Day 1 Cmax) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Accumulation ratio (comparing Day 5 AUCtau to Day 1 AUC0-12) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Area under the plasma-concentration time curve over the first 12 hours after dosing (AUC0-12) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Area under the concentration time curve from time 0 extrapolated to infinity (AUC∞) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Termination elimination half-life (t½) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Apparent total body clearance (CL/F) | Up to 8 days
  Blood Samples will be collected for plasma analysis
PK of AVR-48 in plasma: Apparent volume of distribution during the terminal elimination phase (Vz/F) | Up to 8 days
  Blood Samples will be collected for plasma analysis

CONTACTS AND LOCATIONS:
Overall Officials: Suchismita Acharya, PhD, Study Director — AyuVis Research, Inc.
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No